CLINICAL TRIAL: NCT06810609
Title: Prospective Randomized Phase II Trial on Induction Immunochemotherapy Followed by Surgery or Definitive Chemoradiation and Consolidation Durvalumab (MEDI4736) in Resectable and Borderline Resectable Stage IIIA/B NSCLC
Brief Title: Immunochemotherapy, Surgery or Chemoradiation, and Durvalumab for Stage IIIA/B NSCLC
Acronym: InDuRanS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Eleni Gkika, Prof. Dr. med., University Hospital, Bonn
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESR-21-21565; 2024-516367-80-00 (EU CTIS Number)
Record Dates: First submitted 2025-01-24; First posted 2025-02-05 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-05

CONDITIONS: Lung Cancer Non-Small Cell Cancer (NSCLC)
Keywords: InDuRanS; Non-Small Cell Lung Cancer; Chemoradiation; Resectable NSCLC; Durvalumab; Induction Immunochemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Surgical Procedures, Operative; Chemoradiotherapy; Immunotherapy

STUDY DESIGN:
Intervention Model Description: The study involves randomizing participants to different treatment arms (induction immunochemotherapy, followed by surgery or chemoradiation, and then consolidation Durvalumab immunotherapy), with the goal of comparing the outcomes between those receiving the full treatment regimen and other treatment options.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Surgery + Immunotherapy (Experimental): Surgical removal of metastasis and consolidation Durvalumab immunotherapy.
  Interventions: Procedure: surgery (any volume) and / or pharmaceuticals treatment initiated or planned or only dynamic observation, in accordance with current clinical guidelines; Drug: Immunotherapy
- Chemoradiotherapy + Immunotherapy (Experimental): Chemoradiotherapy (CRT) followed by consolidation immunotherapy with Durvalumab .
  Interventions: Radiation: Chemoradiotherapy; Drug: Immunotherapy

INTERVENTIONS:
Procedure: surgery (any volume) and / or pharmaceuticals treatment initiated or planned or only dynamic observation, in accordance with current clinical guidelines — Surgical removal of the tumor in patients with resectable or borderline resectable NSCLC
  Arms: Surgery + Immunotherapy
Radiation: Chemoradiotherapy — Chemoradiotherapy
  Arms: Chemoradiotherapy + Immunotherapy
Drug: Immunotherapy — Immunotherapy (Durvalumab).

SUMMARY:
The hypothesis of the study is that induction immunochemotherapy, followed by surgery or chemoradiation and consolidation Durvalumab immunotherapy, can significantly improve event-free survival in patients with resectable or borderline resectable NSCLC at stage IIIA/B compared to existing treatment methods.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization (European Union [EU] Data Privacy Directive in the EU) obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.

2. Patient is willing and able to comply with the protocol for the duration of the study 3. Age ≥ 18 years and < 75 years. 4. All sex and gender. 5. Female patients of childbearing potential as well as male patients with partners of childbearing potential must agree to always use a highly effective form of contraception according to the Clinical Trials Facilitation and Coordination Group (CTFG) during the course of this study and for at least 90 days after the last dose of durvalumab or 6 months after the last dose of chemotherapy, whichever occurs last.

6. Evidence of post-menopausal status or negative serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrhoeic for 12 months without an alternative medical cause.

7. Histologically and / or cytologically proven NSCLC (EGFRm-, ALK-). 8.

Selected patients with NSCLC stage IIIA/B:

1. IIIA: one or more lymph node levels involved at EBUS/mediastinoscopy T1/T2 N2.
2. IIIB: one or more lymph node levels involved at EBUS/mediastinoscopy T3/T4 N2. 9. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1. 10. Given technical/oncologic complete resectability (R0) at the time of inclusion. 11. Sufficient functional reserves for the planned surgery 12. Fulfilment of adequate criteria for functional and medical resectability as described in the European Respiratory Society (ERS)/ European Society of Thoracic Surgeons (ESTS) guidelines (Brunelli et al. 2009) and acceptable general clinical condition for multimodality treatment (interdisciplinary committee).

   13. Life expectancy of > 12 weeks. 14. Body weight > 30 kg. 15.

   Adequate normal organ and bone marrow function as defined below:

a. Hemoglobin ≥ 9.0 g/dL. b. Absolute neutrophil count (ANC) ≥ 1.5 × 109/L. c. Platelet count ≥ 100 × 109/L. d. Serum bilirubin ≤ 1.5 × institutional upper limit of normal (ULN). (This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.

e. Alanine aminotransferase (ALT/SGPT) and aspartate aminotransferase (AST/SGOT) ≤ 2.5 × institutional ULN.

f. Measured creatinine clearance (CL) ≥ 60 mL/min or calculated creatinine CL ≥ 60 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance.

16. Stable cardiac function (no myocardial infarction (MI) within 6 months, no heart failure NYHA III-IV).

17. Discussion in a multidisciplinary tumor board which supports participation in this clinical trial, indicating that both chemoradiotherapy and surgery are possible local treatments.

Patients should only be randomized if all of the following inclusion criteria are fulfilled at the time of randomization:

1. Given technical/oncologic complete resectability (R0) at the time of randomization.
2. Sufficient functional reserves for the planned surgery
3. Adequate normal organ and bone marrow function as defined before

   Exclusion Criteria:

1. Unresectable disease. 2. Mixed histology with areas of small cell carcinoma (neuroendocrine markers). 3. ALK+/ EGFRm disease. 4. Clinically symptomatic vena cava superior syndrome. 5. Diffuse mediastinal involvement. 6. Patients with N3 tumors (IASLC/UICC 8). 7. Invasion of the thoracic aorta (T4 - aorta) or the heart (except left atrium - T4 - heart) or the esophagus (T4 - esophagus), or invasion of spine (T4 - spine) NOTE: T4 with invasion of diaphragm are eligible. 8. Pancoast-syndrome in tumors of the superior sulcus (T3-4 Nx). 9. Metastatic disease (M1). 10. Endobronchial tumor extension to the contralateral main stem bronchus. 11. Lung or heart function not allowing the intended surgical procedure at the time of inclusion.

12. Prior treatments including prior mediastinal irradiation. 13. Insufficient patients' compliance (e.g., symptomatic psychiatric disorder) or missing written informed consent or definitive refusal for participation.

14. Prior randomization of treatment in a previous durvalumab clinical study regardless of treatment arm assignment.

15.

Patients who have received prior anti-PD-1, anti-PD-L1, or anti-CTLA-4:

1. Must not have experienced a toxicity that led to permanent discontinuation of prior immunotherapy.
2. All AEs while receiving prior immunotherapy must have completely resolved or resolved to baseline prior to screening for this study.
3. Must not have experienced a ≥ Grade 3 immune related AE or an immune related neurologic or ocular AE of any grade while receiving prior immunotherapy.

   NOTE: Patients with endocrine AE of ≤ Grade 2 are permitted to be enrolled if they are stably maintained on appropriate replacement therapy and are asymptomatic.
4. Must not have required the use of additional immunosuppression other than corticosteroids for the management of an AE, not have experienced recurrence of an AE if re-challenged, and not currently require maintenance doses of > 10 mg prednisone or equivalent per day.

   16. Participation in another clinical study with an investigational product during the last 12 months.

   17. Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.

   18. History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest CT scan.

   19. Any concurrent chemotherapy (other than study therapy), Investigational Product, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.

   20. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of durvalumab.

   21. History of allogenic organ transplantation or a stem cell transplantation. 22.

   Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

a. Vitiligo or alopecia b. Hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement c. Any chronic skin condition that does not require systemic therapy d. Celiac disease controlled by diet alone e. Patients without active disease in the last 5 years may be included but only after consultation with the study physician 23. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.

24. History of another primary malignancy except for

a. Malignancy treated with curative intent and with no known active disease ≥ 5 years before the first dose of durvalumab and of low potential risk for recurrence b. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease c. Adequately treated carcinoma in situ without evidence of disease 25. History of active primary immunodeficiency. 26. History of leptomeningeal carcinomatosis. 27. Known active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B, hepatitis C, or human immunodeficiency virus (positive HIV-1 or HIV-2). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.

28.

Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

1. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
2. Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication) 29. Current or prior use of immunostimulatory agents within 14 days before the first dose of durvalumab 30. Receipt of live attenuated vaccine within 30 days prior to the first dose of durvalumab. Note: Patients, if enrolled, should not receive live vaccine whilst receiving study treatment and up to 90 days after the last dose of study treatment.

   31. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab or 6 months after the last dose of chemotherapy, whichever occurs last.

   32. Known allergy or hypersensitivity to any of the study drugs or any of the study drugs excipient.

   33. Any medical contraindication to treatment with platin-based doublet chemotherapy as listed in the applying SmPCs.

   34. Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.

   Patients should not be randomized if any of the following exclusion criteria are fulfilled at the time of randomization:

   1. Complete remission after induction immunochemotherapy. 2.

   Any unresolved toxicity NCI CTCAE Grade ≥ 2 from previous immunochemotherapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria:

a. Patients with Grade ≥ 2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.

b. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Study Physician (exception: alopecia).

3. Allergy or hypersensitivity to durvalumab or concurrent chemotherapy drugs or any excipient appearing for the first time during previous immunochemotherapy.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2025-04-20 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
2-Year Event-Free Survival (EFS) Rate in Patients with Resectable or Borderline Resectable NSCLC | Within 2 years after date of randomization
  2 year EFS rate is defined as percentage of patients without an event specified as relapse or progression according to RECIST 1.1 criteria, secondary tumor, or death of any cause, whichever occurs first, within 2 years after date of randomization.

SECONDARY OUTCOMES:
Analyze the health-related Quality of Life (QoL) | from date of randomization through study completion (an average of 14 months after randomization)
  Changes in European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) C30 symptom scales from date of randomization through study completion (an average of 14 months after randomization) and changes in EORTC QLQ-C30 functional scales and global health status from date of randomization through study completion (an average of 14 months after randomization). Higher scores indicate a better outcome.
Analyze the health-related Quality of Life (QoL) | from date of randomization through study completion (an average of 14 months after randomization)
  Changes in European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) LC13 symptom scales from date of randomization through study completion (an average of 14 months after randomization). Higher scores indicate a better outcome.
Occurence of adverse events | for 12 months according to arm
  Occurrence of adverse events according to CTCAE (V5.0):
  * adverse events grade ≥ 3 (according to NCI CTCAE v5.0)
  * SAEs
  * Unexpected AEs
Efficacy of multimodality treatment | From Randomization to death from any cause, within 2 years after date of randomization or throughout extended follow-up
  Efficacy will be assessed in terms of Overall survival (OS) defined as time from randomization until death due to any cause
Efficacy of multimodality treatment | From Randomization to objective disease progression, within 2 years after date of randomization or throughout extended follow-up
  Efficacy will be assessed in terms of Progression free survival (PFS) defined as time from randomization to objective disease progression
Outcome of surgery in resected patients | end of surgery
  Assessment of rate of pathological complete response (pCR), major pathological response (mPR) and R0 in resected patients
Response after induction therapy | pre-induction therapy scan in comparison with post-induction therapy scan
  Assessment of Functional response (FDG-PET-CT-scan) to induction therapy prior to thoracotomy / chemoradiation according to RECIST and PERCIST in the whole population and in both arms according to CR, PR, SD and PD
Response after induction therapy | pre-induction therapy scan in comparison with post-induction therapy scan
  Analysis of the SUVmax response and MTV response on the planning FDG-PET-CT in comparison to the pretreatment FDG-PET-CT
Quantity of PD-L1 positive tumor cells per patient | At screening visit
  Assessment of number of PD-L1 positive tumor cells at screening visit.
Rate of patients with < 1%, 1-49% and ≥ 50 % PD-L1 positive tumor cells in the group of stage IIIA/B (N2) NSCLC patients (screened population), | From Screening
  Assessment of the rate of patients with < 1%, 1-49% and ≥ 50 % PD-L1 positive tumor cells in the group of stage IIIA/B (N2) NSCLC patients (screened population).
Compliance and treatment toxicity effects | From randomization until end of treatment visit, an average of 14 months after randomization
  Assessment of Rate of randomized patients who completed the planned treatment
Compliance and treatment toxicity effects | From randomization until end of treatment visit, an average of 14 months after randomization
  Assessment of Rate of patients who discontinued study treatment due to adverse event
Toxicity of ICT and any causes that prevent randomization or surgery or completion of surgery | Before Randomization
  Assessment of rate of patients with events / PD that prevent fulfillment of criteria for randomization / surgery

OTHER OUTCOMES:
Radiological response including radiomics in irradiated patients. | from randomization into arm 2 (chemoradiotherapy) till study completion (an average of 14 months after randomization) or throughout extended follow-up
  Assessment of correlation of radiomic features with the treatment response (only for patients in the chemoradiation arm)
Training and evaluation of deep learning algorithms for automated response prediction | from enrollment till study completion (an average of 17 months after enrollment) or throughout extended follow-up
  compared with physician-assessed response evaluation
Training and evaluation of deep learning algorithms for automated assessment of Tumor Progression Patterns | from enrollment till study completion (an average of 17 months after enrollment) or throughout extended follow-up
  compared with physician-assessed Tumor Progression Patterns
Assessment of blood samples for ctDNA and plasma proteomics | from enrollment till study completion (an average of 17 months after enrollment) or throughout extended follow-up
  Assessment of amount of ctDNA and further analysis including sequencing, characterization and quantification of plasma proteins
Immune responses | from enrollment till study completion (an average of 17 months after enrollment) or throughout extended follow-up
  Immunoprofiling of peripheral blood cells using flow cytometry

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (5):
  - University Hospital Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Klinikum Stuttgart, Stuttgart, Baden-Wurttemberg
  - University Hospital Gießen, Giessen, Hesse
  - Johannes Wesling Klinikum Minden Mühlenkreiskliniken, Hämatologie und Onkologie, Minden, North Rhine-Westphalia
  - University Hospital Bonn, Bonn